CLINICAL TRIAL: NCT05085834
Title: Zinc Effect on Inflammation and Cardiovascular Risk in HIV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Grace McComsey, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Zinc study; 1R21AT009153 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2021-10-20 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Inflammation; Cardiovascular Diseases; Zinc Deficiency
Keywords: Zinc; inflammation; Cardiovascular Diseases risk
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases | interventions — gluconic acid

STUDY DESIGN:
Intervention Model Description: This is a double-blind randomized placebo-controlled trial 2:1 Patients will be given zinc gluconate capsules at a dose of 90 mg elemental zinc daily or matching placebo for 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, study staff, and the study statistician will be blinded to treatment allocation (zinc gluconate or placebo capsules). The research staff as well as the principle investigator will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zinc gluconate (Experimental): Patients received Zinc gluconate 45 mg capsules orally twice daily for 24 weeks.
  Interventions: Drug: Zinc Gluconate
- Placebo (Placebo Comparator): Patients received Zinc gluconate Placebo capsules orally twice daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc Gluconate — Two 45 mg capsules once daily
  Arms: Zinc gluconate
Drug: Placebo — Two placebo capsules once daily
  Arms: Placebo

SUMMARY:
To study the effect of short-term zinc supplementation on improving inflammation, metabolic, and cardiovascular risk among HIV infected patients on stable anti-retroviral therapy

DETAILED DESCRIPTION:
This study will focus on subjects with documented zinc deficiency (levels <75 µg/dl) as group most likely to benefit from the zinc supplementation. The investigators also acknowledge that zinc may be beneficial in all HIV subjects, regardless of the plasma zinc level; however initial studies should be done in subjects with low zinc levels as they are more likely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Documentation of an HIV-1 RNA level of ≤400 copies/mL in the last 4 months prior to study entry
* Male or Female age ≥18 years
* Zinc level ≤0.75 mg/L in the last 60 days

Exclusion Criteria:

* Pregnancy/lactation
* Known cardiovascular disease
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace A McComsey, MD, FIDSA, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zinc Gluconate | Placebo
Started | 63 | 32
Completed | 47 | 29
Not Completed | 16 | 3
Not completed — Lost to Follow-up | 9 | 2
Not completed — Adverse Event | 6 | 0
Not completed — Death | 1 | 0
Not completed — Inability to swallow the pill | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc Gluconate | Placebo | Total
Number analyzed (Participants) | 63 | 32 | 95
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.42 [38.92 to 60.55] | 53.29 [45.31 to 58.90] | 52.42 [40.34 to 60.12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 6 | 25
  Male | 44 | 26 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 57 | 27 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 18 | 56
  White | 23 | 14 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
alcohol (current) [Count of Participants; unit: Participants] | 45 | 21 | 66
smokers (current) [Count of Participants; unit: Participants] | 16 | 13 | 29
CD4+ T-Cell Count [Median (Inter-Quartile Range); unit: cells/mm³] | 747.00 [529.00 to 1024.00] | 668.00 [507.00 to 775.00] | 722.00 [526.00 to 973.00]
HIV RNA (<20 copies) [Count of Participants; unit: Participants] | 51 | 23 | 74
Anti-Retroviral Treatment Duration [Median (Inter-Quartile Range); unit: Months] | 178.76 [107.20 to 232.51] | 167.86 [115.14 to 239.51] | 171.86 [108.22 to 236.36]
Protease Inhibitor use [Count of Participants; unit: Participants] | 8 | 7 | 15
Body Mass Index BMI [Median (Inter-Quartile Range); unit: kg/m2] | 28.34 [24.80 to 32.70] | 27.45 [23.23 to 32.40] | 28.08 [24.62 to 32.70]
Waist circumference [Median (Inter-Quartile Range); unit: cm] | 96.67 [89.83 to 106.33] | 97.83 [87.50 to 106.42] | 97.00 [89.17 to 106.33]
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 125 [117 to 139] | 129 [118.5 to 141] | 126 [117 to 141]
Diastolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 80 [75 to 85] | 82 [77 to 88.5] | 81 [75 to 86]
Non-High Density Lipoprotein non-HDL cholesterol [Median (Inter-Quartile Range); unit: (mg/dL] | 115.30 [98 to 147.6] | 115.50 [93.90 to 166.25] | 115.30 [95.7 to 149.2]
High Density Lipoprotein [Median (Inter-Quartile Range); unit: mg/dL] | 45.40 [39.80 to 60.80] | 48.15 [41.30 to 62.70] | 47.00 [39.90 to 61.10]
Low Density Lipoprotein LDL [Median (Inter-Quartile Range); unit: mg/dl] | 96 [74 to 114] | 89 [66.5 to 127.5] | 96 [71 to 118]
Very Low Density Lipoprotein VLDL [Median (Inter-Quartile Range); unit: mg/dl] | 22 [15 to 29] | 20 [15 to 27] | 21 [15 to 28.5]
Cholesterol [Median (Inter-Quartile Range); unit: mg/dl] | 171 [144 to 192] | 165.5 [147.5 to 213.5] | 169 [144 to 202]
cholesterol/ high Density Lipoprotein Ratio [Median (Inter-Quartile Range); unit: Ratio] | 3.5 [2.8 to 4.4] | 3.2 [2.55 to 4.85] | 3.4 [2.7 to 4.4]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dl] | 108 [71 to 146] | 103 [76.5 to 136] | 105 [74 to 146]
Insulin [Median (Inter-Quartile Range); unit: mIU/mL] | 10 [6 to 17] | 11.5 [6.5 to 18.5] | 10.5 [6 to 18]
atherosclerotic cardiovascular risk 10 year ASCVD [Median (Inter-Quartile Range); unit: %] — probability (%) that an individual will have a first major ASCVD event (like a heart attack or stroke) within the next 10 years.
  % | 6.1 [2.7 to 11.1] | 6.7 [3.85 to 12.5] | 6.5 [2.9 to 11.8]
Presence of metabolic syndrome [Count of Participants; unit: Participants] | 26 | 14 | 40
Endothelial Function: Reactive Hyperemic Index [Median (Inter-Quartile Range); unit: ratio] — Endothelial function was assessed noninvasively using RH-PAT (EndoPAT 2000) with finger probes and brachial occlusion-induced hyperemia.
  A Reactive Hyperemia Index (RHI) was calculated from the change in pulse wave amplitude (PWA) relative to the pulse wave amplitude (PWA) before the occlusion of the artery, in the occluded arm, corrected for corresponding changes in the contralateral, non-occluded arm to minimize the influence of non-endothelial-dependent systemic effects. An RHI value greater than 1.67 is considered normal. Higher values indicate better endothelial function.
  ratio | 1.91 [1.6 to 2.21] | 1.89 [1.62 to 2.04] | 1.9 [1.6 to 2.19]
Endothelial Function: Augmentation Index [Median (Inter-Quartile Range); unit: %] | 7.5 [-2 to 14] | 11 [4 to 16] | 10 [-1 to 15]
hsCRP [Median (Inter-Quartile Range); unit: ng/mL] | 2240.00 [1075.40 to 7930.31] | 1998.85 [967.08 to 6778.08] | 2202.14 [993.51 to 7795.00]
sCD14 [Median (Inter-Quartile Range); unit: ng/mL] | 1671.20 [1424.41 to 2001.68] | 1727.05 [1525.77 to 1963.90] | 1681.63 [1468.60 to 1966.05]
sCD163 [Median (Inter-Quartile Range); unit: ng/mL] | 543.40 [366.03 to 778.58] | 593.61 [461.03 to 784.74] | 568.55 [420.62 to 780.63]
sTNFR-I [Median (Inter-Quartile Range); unit: pg/mL] | 1036.85 [890.50 to 1183.57] | 977.39 [819.30 to 1200.68] | 1006.42 [881.12 to 1195.08]
sTNFR-II [Median (Inter-Quartile Range); unit: pg/mL] | 2162.27 [1889.96 to 2867.83] | 2253.23 [1923.78 to 3031.33] | 2234.54 [1907.77 to 2912.41]
DDimer [Median (Inter-Quartile Range); unit: ng/mL] | 558.43 [389.36 to 883.46] | 520.93 [293.47 to 717.11] | 536.22 [366.79 to 809.72]
oxLDL [Median (Inter-Quartile Range); unit: U/L] | 51731.12 [41091.65 to 75262.57] | 47606.57 [37342.25 to 62313.38] | 50145.48 [39945.47 to 70630.87]
IL-6 [Median (Inter-Quartile Range); unit: pg/mL] | 2.11 [1.26 to 3.46] | 1.89 [1.42 to 3.51] | 1.94 [1.31 to 3.46]
VCAM [Median (Inter-Quartile Range); unit: ng/mL] | 758.04 [658.95 to 950.49] | 857.01 [693.53 to 1013.78] | 783.99 [671.49 to 970.46]
ICAM [Median (Inter-Quartile Range); unit: ng/mL] | 244.28 [180.09 to 298.24] | 250.13 [175.81 to 290.17] | 247.37 [180.09 to 293.93]
IP-10 [Median (Inter-Quartile Range); unit: pg/mL] | 130.52 [102.35 to 207.19] | 134.70 [90.04 to 190.78] | 134.48 [99.61 to 199.31]
LBP [Median (Inter-Quartile Range); unit: μg/mL] | 16.6 [13.16 to 30.47] | 16.44 [12.55 to 20.35] | 16.6 [12.77 to 25.77]
IFAB [Median (Inter-Quartile Range); unit: pg/mL] | 1826.49 [1131.22 to 2741.16] | 1616.94 [996.70 to 2295.69] | 1730.93 [1087.46 to 2681.82]
BDG [Median (Inter-Quartile Range); unit: pg/mL] | 98.46 [72.89 to 164.33] | 122.51 [87.07 to 197.11] | 106.08 [77.72 to 168.20]
Zonulin [Median (Inter-Quartile Range); unit: μg/mL] | 1020 [674.68 to 1390] | 1040 [665.92 to 1460] | 1030 [674.68 to 1440]
Zinc level [Median (Inter-Quartile Range); unit: μg/dL] | 70 [66 to 72.2] | 69 [61.2 to 73] | 69.8 [64.3 to 73]

OUTCOME MEASURES:

1. Primary Outcome: Effect of Zinc Supplementation on Zinc Levels at 24 Weeks in HIV-infected Subjects
Description: Changes in zinc levels after zinc supplementation in HIV-infected subjects with zinc deficiency
Time Frame: between baseline and 24 weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: absolute change (μg/dL)
Groups:
- Placebo: participants assigned to the placebo group
- Zinc 90 mg: participants assigned to the Zinc group
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
absolute change (μg/dL) | 8.60 [1.65 to 20.00] | 33.50 [14.00 to 62.70]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Zinc, μg/dL); Test type: Other — Generalized estimating equations were used while adjusting for age and sex, and examining interactions between time and treatment. Combining linear coefficients in the equation while accounting for the multiplicative effects of treatment and time were considered to assess the true effect size of zinc supplementation on biomarkers; p < 0.01, linear combination of coefficients; β coefficient = 0.71, 95% CI 2-sided [0.43 to 0.98], Standard Error of Mean 0.14

2. Primary Outcome: Effect of Zinc Supplementation on Inflammation and Immune Activation in HIV-infected Subjects
Description: Changes in markers of inflammation and immune activation by measuring monocyte activation soluble markers CD14 (sCD14), and soluble CD163 (sCD163), high sensitivity C reactive protein (hsCRP), D-dimer, vascular cell adhesion molecule-1 (VCAM), and intercellular adhesion molecule-1 (I-CAM)
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
ng/mL
  hsCRP (ng/mL) | -22.86 [-689.27 to 1744.48] | 1.33 [-602.56 to 1174.87]
  sCD14 (ng/mL) | 101.71 [-90.50 to 243.20] | -56.31 [-263.24 to 134.19]
  sCD163 (ng/mL) | -50.11 [-153.06 to 89.80] | 43.69 [-102.27 to 126.91]
  D-dimer (ng/mL) | -149.05 [-294.46 to 58.72] | -45.85 [-295.57 to 142.43]
  VCAM (ng/mL) | 66.69 [-2.65 to 187.38] | 49.53 [-55.61 to 170.15]
  ICAM (ng/mL) | -2.03 [-28.37 to 22.30] | 2.35 [-29.19 to 42.46]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(hsCRP ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 1.00, linear combination of coefficients; β coefficient = -0.002, 95% CI 2-sided [-0.57 to 0.57], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(sCD14, ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.08, linear combination of coefficients; β coefficient = -0.08, 95% CI 2-sided [-0.18 to 0.01], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(sCD163, ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.77, linear combination of coefficients; β coefficient = -0.03, 95% CI 2-sided [-0.21 to 0.15], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(D-dimer, ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.19, linear combination of coefficients; β coefficient = 0.2, 95% CI 2-sided [-0.10 to 0.50], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(VCAM, ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.10, linear combination of coefficients; β coefficient = -0.19, 95% CI 2-sided [-0.41 to 0.04], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(ICAM, ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.98, linear combination of coefficients; β coefficient = 0.41, 95% CI 2-sided [-39.16 to 39.98], Standard Error of Mean 20.19

3. Primary Outcome: Effect of Zinc Supplementation on Inflammation in HIV-infected Subjects
Description: Changes in markers of inflammation and immune activation by measuring soluble tumor necrosis alpha receptor I and II (sTNFR-I and II), Interleukin-6 (IL-6), and interferon-gamma-inducible protein of 10 kDa (IP-10).
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
pg/mL
  sTNF-RI (pg/mL) | -25.08 [-209.51 to 186.66] | 1.27 [-236.80 to 168.27]
  sTNF-RII (pg/mL) | -121.65 [-457.93 to 467.29] | 99.33 [-484.31 to 477.72]
  IL-6 (pg/mL) | -0.47 [-0.85 to 0.61] | -0.02 [-0.88 to 0.72]
  IP-10 (pg/mL) | 0.23 [-44.28 to 29.08] | -9.99 [-31.65 to 20.27]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(sTNF-RI , pg/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.55, linear combination of coefficients; β coefficient = 0.04, 95% CI 2-sided [-0.09 to 0.16], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(sTNF-RII, pg/m); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.95, linear combination of coefficients; β coefficient = -0.004, 95% CI 2-sided [-0.13 to 0.13], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(IL-6, pg/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.73, linear combination of coefficients; β coefficient = 0.07, 95% CI 2-sided [-0.30 to 0.43], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(IP-10, pg/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.48, linear combination of coefficients; β coefficient = 0.12, 95% CI 2-sided [-0.22 to 0.47], Standard Error of Mean 0.18

4. Primary Outcome: Effect of Zinc on oxLDL in HIV-infected Subjects
Description: Changes in oxidized low density lipoprotein (OxLDL) (U/L) over 24 weeks
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
U/L | 20833.33 [2397.72 to 61644.46] | 8639.79 [-1716.35 to 43693.14]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(OxLDL, U/L); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.83, linear combination of coefficients; β coefficient = 1819.18, 95% CI 2-sided [-14899.37 to 18537.74], Standard Error of Mean 8530.03

5. Secondary Outcome: Effect of Zinc Supplementation on Metabolic Markers at 24 Weeks in HIV-infected Subjects
Description: Changes in metabolic markers after zinc supplementation by measuring Non-HDL cholesterol, high-density lipoprotein (HDL), low density lipoprotein (LDL), very low density lipoprotein (VLDL), Cholesterol, Cholesterol - HDL Ratio, and Triglycerides.
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
mg/dL
  Non-HDL cholesterol (mg/dL) | 3.10 [-28.20 to 26.50] | 1.35 [-12.30 to 10.85]
  HDL (mg/dL) | -1.70 [-4.60 to 1.40] | -2.45 [-8.45 to 1.25]
  LDL (mg/dL) | 6.00 [-28.00 to 16.00] | -1.50 [-19.50 to 11.50]
  VLDL (mg/dL) | 0.50 [-6.00 to 3.50] | 2.00 [-2.00 to 6.00]
  Cholesterol (mg/dL) | 2.00 [-25.00 to 27.00] | -3.50 [-23.50 to 12.00]
  Triglycerides (mg/dL) | 2.00 [-29.00 to 12.00] | 7.00 [-12.50 to 34.50]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Non-HDL Cholesterol (mg/dL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.84, linear combination of coefficients; β coefficient = 0.01, 95% CI 2-sided [-0.12 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(HDL (mg/dL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.18, linear combination of coefficients; β coefficient = -0.08, 95% CI 2-sided [-0.19 to 0.04], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(LDL (mg/dL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.84, linear combination of coefficients; β coefficient = -0.02, 95% CI 2-sided [-0.19 to 0.15], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(VLDL (mg/dL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.55, linear combination of coefficients; β coefficient = 0.07, 95% CI 2-sided [-0.15 to 0.29], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Cholesterol (mg/dl)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.78, linear combination of coefficients; β coefficient = -0.01, 95% CI 2-sided [-0.11 to 0.09], Standard Error of Mean 0.05
Statistical Analysis 6: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Triglycerides (mg/dL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.58, linear combination of coefficients; β coefficient = 0.07, 95% CI 2-sided [-0.17 to 0.31], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on Metabolic Syndrome; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.35, linear combination of coefficients; β coefficient = -0.44, 95% CI 2-sided [-1.36 to 0.48], Standard Error of Mean 0.47

6. Secondary Outcome: Effect of Zinc Supplementation on Cholesterol - HDL Ratio at 24 Weeks in HIV-infected Subjects
Description: Changes in metabolic markers after zinc supplementation for 24 weeks by measuring the Cholesterol - HDL Ratio
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
Ratio | 0.10 [-0.20 to 0.40] | 0.10 [-0.10 to 0.45]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Chol:HDL Ratio); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.36, linear combination of coefficients; β coefficient = 0.06, 95% CI 2-sided [-0.07 to 0.20], Standard Error of Mean 0.07

7. Secondary Outcome: the Effect of Zinc Supplementation on BMI at 24 Weeks in HIV-infected Subjects
Description: Changes in metabolic markers after zinc supplementation by measuring the body mass index (BMI) (kg/m2)
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: kg/m2
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
kg/m2 | 0.28 [-0.52 to 1.16] | 0.10 [-0.58 to 0.95]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on BMI (kg/m2); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.86, linear combination of coefficients; β coefficient = -0.35, 95% CI 2-sided [-4.29 to 3.60], Standard Error of Mean 2.01

8. Secondary Outcome: Effect of Zinc on the Waist-umbilicus at 24 Weeks in HIV-infected Subjects
Description: Changes in metabolic markers after zinc supplementation by measuring Waist-umbilicus (cm)
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
cm | 0.50 [-2.53 to 2.50] | 1.67 [-2.67 to 3.00]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Waist-umbilicus (cm)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.74, linear combination of coefficients; β coefficient = -0.01, 95% CI 2-sided [-0.08 to 0.05], Standard Error of Mean 0.03

9. Secondary Outcome: Effect of Zinc Supplementation on Weight at 24 Weeks in HIV-infected Subjects
Description: Changes in metabolic markers after zinc supplementation by measuring body weight (lbs)
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: lbs
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
lbs | 2.20 [-3.50 to 7.60] | 0.00 [-4.00 to 4.40]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on Weight (lbs); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.81, linear combination of coefficients; β coefficient = -2.99, 95% CI 2-sided [-26.97 to 20.99], Standard Error of Mean 12.23

10. Secondary Outcome: Effect of Zinc Supplementation on Blood Pressure at 24 Weeks in HIV-
Description: Changes in metabolic markers after zinc supplementation by measuring Systolic Blood Pressure and Diastolic Blood Pressure (mmHg)
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
mmHg
  Systolic Blood Pressure (mmHg) | 6.00 [-4.00 to 12.00] | 0.00 [-9.00 to 9.00]
  Diastolic Blood Pressure (mmHg) | 3.00 [-5.00 to 6.00] | 0.00 [-5.00 to 5.00]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Systolic blood pressure (mmHg)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.41, linear combination of coefficients; β coefficient = -0.02, 95% CI 2-sided [-0.07 to 0.03], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on Diastolic blood pressure (mmHg); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.42, linear combination of coeff; β coefficient = -1.68, 95% CI 2-sided [-5.71 to 2.36], Standard Error of Mean 2.06

11. Secondary Outcome: Effect of Zinc Supplementation on 10 Year Atherosclerotic Cardiovascular Disease at 24 Weeks in HIV-infected Subjects
Description: Changes in metabolic markers after zinc supplementation were measured by measuring 10-year atherosclerotic cardiovascular disease (ASCVD), which is the probability (%) that an individual will have a first major ASCVD event (like a heart attack or stroke) within the next 10 years with higher scores indicating worse outcome
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: percentage of 10-year ASCVD score
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
percentage of 10-year ASCVD score | 0.40 [-1.10 to 2.00] | 0.00 [-1.35 to 1.55]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(10 year ASCVD (%)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.70, linear combination of coefficients; β coefficient = -0.04, 95% CI 2-sided [-0.26 to 0.17], Standard Error of Mean 0.11

12. Secondary Outcome: Effect of Zinc Supplementation on Endothelial Function in HIV-infected Subjects
Description: Changes in markers of endothelial function including the Reactive Hyperemic Index and Augmentation Index Endothelial function was assessed noninvasively using RH-PAT (EndoPAT 2000) with finger probes and brachial occlusion-induced hyperemia.
  A Reactive Hyperemia Index (RHI) was calculated from the change in pulse wave amplitude (PWA) relative to baseline in the occluded arm, corrected for corresponding changes in the contralateral, non-occluded arm to minimize the influence of non-endothelial-dependent systemic effects. An RHI value greater than 1.67 is considered normal, while a value of 1.67 or lower is considered abnormal. Higher values indicate better endothelial function.
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: (ratio) absolute change
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
(ratio) absolute change
  Reactive Hyperemic Index | -0.34 [-0.77 to 0.16] | -0.18 [-0.60 to 0.23]
  Augmentation Index | 0.00 [-8.00 to 5.50] | -1.00 [-7.00 to 6.00]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on Reactive Hyperemic Index; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.62, linear combination of coefficients; β coefficient = -0.03, 95% CI 2-sided [-0.17 to 0.10], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on Augmentation Index; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.81, linear combination of coefficients; β coefficient = 0.59, 95% CI 2-sided [-4.19 to 5.36], Standard Error of Mean 2.43

13. Secondary Outcome: Effect of Zinc Supplementation on IFAB and BDG in HIV-infected Subjects
Description: Changes in markers of Gut Integrity Markers including: intestinal fatty acid-binding protein (IFAB) and (1,3)-β-d-glucan (BDG)
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
pg/mL
  IFAB (pg/mL) | 100.82 [-747 to 953.32] | 58.89 [-1049.29 to 654.96]
  BDG (pg/mL) | -28.19 [-100.43 to 4.02] | 8.36 [-63.26 to 76.12]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(IFAB (pg/mL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.90, linear combination of coefficients; β coefficient = 0.02, 95% CI 2-sided [-0.26 to 0.30], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(BDG (pg/mL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.24, linear combination of coefficients; β coefficient = 0.18, 95% CI 2-sided [-0.12 to 0.47], Standard Error of Mean 0.15

14. Secondary Outcome: Effect of Zinc Supplementation on LBP and Zonuline in HIV-infected Subjects
Description: Changes in markers of Gut Integrity Markers including: lipopolysaccharide-binding protein (LBP) and Zonulin.
Time Frame: between baseline and 24 Weeks
Population: absolute changes for outcome measures over 24 weeks for each group
Measure: Median (Inter-Quartile Range); unit: μg/mL
Arm/Group | Placebo | Zinc 90 mg
Number analyzed (Participants) | 32 | 63
μg/mL
  LBP (μg/mL) | 0.47 [-4.8 to 8.35] | 0.72 [-4.52 to 6.9]
  Zonulin (μg/mL) | 78.2 [-138 to 506.86] | 270.54 [59.36 to 600.45]
Statistical Analysis 1: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(LBP (ng/mL)); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.69, v; β coefficient = 0.05, 95% CI 2-sided [-0.21 to 0.32], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Zinc 90 mg; effect of Zinc supplementation on ln(Zonulin (ng/mL); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.49, linear combination of coefficients; β coefficient = 0.09, 95% CI 2-sided [-0.16 to 0.34], Standard Error of Mean 0.13

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Zinc Gluconate | Placebo
All-Cause Mortality (participants affected / at risk) | 1/63 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/32
Other Adverse Events (participants affected / at risk) | 48/63 | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zinc Gluconate (N=63) | Placebo (N=32)
Death (Injury, poisoning and procedural complications) | 1 | 0 — Death occurred secondary to drug overdose not related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zinc Gluconate (N=63) | Placebo (N=32)
Abdominal adhesions with intestinal torsion (Gastrointestinal disorders) | 1 | 0
Abcess post root canal (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
High Blood Pressure (Cardiac disorders) | 0 | 1
Chest Pain (Cardiac disorders) | 1 | 0
Left groin hernia (Gastrointestinal disorders) | 1 | 0
Pain in right hip and Sciatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral Neuropathy (Nervous system disorders) | 1 | 0
Scrotal Abcess (Skin and subcutaneous tissue disorders) | 0 | 1
Worsening of depression (Psychiatric disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 8 | 0
Stomach Pain (Gastrointestinal disorders) | 2 | 0
High ALT and/or AST (Hepatobiliary disorders) | 8 | 1
High Cholesterol (Metabolism and nutrition disorders) | 14 | 13
High Creatine Kinase (Musculoskeletal and connective tissue disorders) | 6 | 1
High Creatinine (Renal and urinary disorders) | 19 | 17
Low Hemoglobin (Blood and lymphatic system disorders) | 2 | 1
Low Phosphorus (General disorders) | 1 | 2
Low Sodium (General disorders) | 2 | 1
High Sodium (General disorders) | 0 | 1
High Alkaline Phosphatase (Hepatobiliary disorders) | 2 | 0
High Bilirubin (Hepatobiliary disorders) | 2 | 5
High Glucose (Metabolism and nutrition disorders) | 30 | 17
High LDL (Metabolism and nutrition disorders) | 10 | 8
High Triglycerides (Metabolism and nutrition disorders) | 25 | 11
High Uric Acid (Metabolism and nutrition disorders) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT05085834/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT05085834/ICF_001.pdf